

Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Comparative Study and a Phase 3, Multicenter, Open-Label, Long-term Study to Evaluate the Efficacy and Safety of SYR-472 When Orally Administered at a Dose of 25 mg Once Weekly in Patients with Type 2 Diabetes Mellitus Complicated by Severe Renal Impairment or End-Stage Renal Failure

NCT Number: NCT02512068

Statistical analysis plan Approve Date: 19-Jun-2018

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version was Japanese.

# STATISTICAL ANALYSIS PLAN

Study Title : A Phase 3, Multicenter, Randomized, Double-Blind,

Placebo-Controlled, Parallel-Group, Comparative Study and a Phase 3, Multicenter, Open-Label, Long-term Study to Evaluate the Efficacy and Safety of SYR-472 When Orally Administered at a Dose of 25 mg Once Weekly in Patients with Type 2 Diabetes Mellitus Complicated by Severe Renal Impairment or End-Stage

Renal Failure

Protocol No. : SYR-472-3003

Sponsor : Takeda Pharmaceutical Company Limited

| Person responsible for preparing the pro | tocol |
|---|---|
| PPD Ta | keda Pharmaceutical Company Limited |
| PPD | |
| Trial Statistician PPD | Takeda Pharmaceutical Company Limited |
| PPD | |
| PPD | |

Second Version: 19 June 2018

## TABLE OF CONTENTS

| LIST OF ABBREVIATIONS AND DEFINITION OF TERMS | 3 |
|--------------------------------------------------------------------|----|
| HANDLING OF TIME WINDOW | 4 |
| OTHER HANDLING | 11 |
| 1 STUDY SUBJECTS, DEMOGRAPHICS, AND OTHER BASELINE CHARACTERISTICS | 12 |
| 1.1 Disposition of Subjects | 12 |
| 1.1.1 Study Information | 12 |
| 1.1.2 Disposition of All Subjects Who Were Not Randomized | 12 |
| 1.1.3 Subject Eligibility | 12 |
| 1.1.4 Number of Subjects Who Were Randomized by Site | 13 |
| 1.1.5 Disposition of Subjects | 13 |
| 1.1.6 Study Drug Completion Status | 15 |
| 1.1.7 Protocol Deviations and Analysis Sets | 15 |
| 1.2 Demographic and Other Baseline Characteristics. | 16 |
| 1.2.1 Distribution of Baseline Demographics | 16 |
| 1.2.2 Medical History and Concurrent Medical Conditions | 18 |
| 1.2.3 Medication History and Concomitant Medications | 18 |
| 1.2.4 Concomitant Antidiabetic Drugs Permitted in the Study | 19 |
| 1.3 Measurement of Compliance Status for Treatment | 20 |
| 1.3.1 Study Drug Exposure and Compliance in the Treatment Period | 20 |
| 1.3.2 Compliance of Antidiabetic Drugs | 21 |
| 1.3.3 Compliance of Diet and/or Exercise Therapy | 21 |
| 2 EFFICACY ANALYSIS | 22 |
| 2.1 Primary Endpoints and Analysis Methodology | 22 |
| 2.1.1 Primary Analysis | 22 |
| 2.1.2 Secondary Analysis | 22 |
| 2.2 Secondary Endpoints and Analysis Methodology | 23 |
| 2.2.1 HbA1c, Fasting Blood Glucose, Glycoalbumin | 23 |
| 2.3 Other Endpoints and Analysis Methodology | 24 |
| 2.3.1 Fasting C-peptide, Fasting Glucagon, DPP-4 Activity, Weight | 24 |
| 2.4 Statistical and Analytical Issues | 25 |
| 2.4.1 Adjustments for Covariates | 25 |
| 2.4.2 Handling of Dropouts or Missing Data | 25 |
| 2.4.3 Interim Analysis and Data Monitoring | |
| 2.4.4 Multicenter Studies | 25 |
| 2.4.5 Multiple Comparisons/Multiplicity | 25 |
| 2.4.6 Use of an "Efficacy Subset of Subjects" | 25 |

| 2.4.7 Active-Control Studies Intended to Show Equivalence or Non-inferiority | 26 |
|---|---|
| 2.4.8 Examination of Subgroups | 26 |
| 2.5 Plasma Concentration of SYR-472Z. | 27 |
| 3 SAFETY ANALYSIS | 28 |
| 3.1 Treatment-Emergent Adverse Event | 28 |
| 3.1.1 Overview of Treatment-Emergent Adverse Events | 28 |
| 3.1.2 Displays of Treatment-Emergent Adverse Events | 29 |
| 3.1.3 Subgroup Analysis of Treatment-Emergent Adverse Events | 31 |
| 3.2 Pretreatment Event | 32 |
| 3.2.1 Display of Pretreatment Events | 32 |
| 3.3 Clinical Laboratory Evaluations and Other Safety Endpoints | 33 |
| 3.3.1 Clinical Laboratory Evaluations | 33 |
| 3.3.2 Vital Signs, Physical Examination, and Other Observation Items Related to Safety | 34 |
| 4 SIGNIFICANCE LEVEL AND CONFIDENCE COEFFICIENT | 37 |
| History of Revision (version management) | 38 |
| [Appendix 1] SYR-472-3003 Comparison Table for Changes | 1 |

#### LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

- Study Day: The day before the start of the study drug administration will be defined as Day -1 and the day of the start of the study drug administration will be defined as Day 1.
- Follow-up Day for Treatment Period I: The day after the last administration of the study drug for Treatment Period I will be defined as Follow-up Day 1 for Treatment Period I.
- Study Day for Treatment Period II: The day before the start of the study drug administration for Treatment Period II will be defined as Day -1 for Treatment Period II and the day of the start of the study drug administration for Treatment Period II will be defined as Day 1 for Treatment Period II.
- Study Day for SYR-472 25 mg tablet: The day before the start of SYR-472 25 mg tablet will be defined as Day -1 for SYR-472 25 mg tablet and the day of the start of SYR-472 25 mg tablet will be defined as Day 1 for SYR-472 25 mg tablet.
- Follow-up Day for SYR-472 25 mg tablet: The day after the last administration of SYR-472 25 mg tablet will be defined as Follow-up Day 1 for SYR-472 25 mg tablet.
- Treatment groups: SYR-472 25 mg group (subjects who received SYR-472 25 mg in both Treatment Periods I and II), placebo group (subjects who received placebo in Treatment Period I and SYR-472 25 mg in Treatment Period II).
  In this statistical analysis plan (hereinafter referred to as SAP), the treatment groups will be presented as the SYR-472 25 mg/SYR-472 25 mg group and the placebo/SYR-472 25 mg group.
- Summary statistics: number of subjects, mean, standard deviation, maximum, minimum, and quartiles
- Reason for not being treated with the study drug for Treatment Period II: If the subject is "Not
  treated" with the study drug for Treatment Period II, the reason why the administration of study
  drug was discontinued will be analyzed as the reason for not being treated with the study drug
  for Treatment Period II.
- Treatment-emergent adverse event (TEAE): An adverse event whose date of onset occurs on or after the start of the study drug administration. Since there is a possibility that the evaluation result of an adverse event may differ before and after the start of the study drug administration for Treatment Period II, the evaluation result of adverse event to be used for analysis will be defined according to the rules below:
  - > TEAEs that occur before the start of the study drug for Treatment Period II: The analysis will be performed based on the evaluation result entered in the CRF under "Pretreatment Event/Adverse Event (Period 1)."
  - > TEAEs that occur after the start of SYR-472 25 mg tablet: The analysis will be performed based on the evaluation results entered in the CRFs under "Pretreatment Event/Adverse Event (Period 1)" and "Pretreatment Event/Adverse Event (Period 2 and thereafter)." If the

evaluation results differ between "Pretreatment Event/Adverse Event (Period 1)" and "Pretreatment Event/Adverse Event (Period 2 and thereafter)," the evaluation result of "Pretreatment Event/Adverse Event (Period 2 and thereafter)" will be preferentially used.

- Time of onset: In the analysis of TEAEs that occur before the start of the study drug for Treatment Period II, the time of onset will be calculated by defining the day of the start of the study drug administration as day 1. In the analysis of TEAEs that occur after the start of SYR-472 25 mg tablet, it will be calculated by defining the day of the start of SYR-472 25 mg tablet as day 1.
- Number of days from the immediate study drug administration: To be calculated by defining the day of the immediate study drug administration as Day 1. If the study drug administration and TEAE occur on the same day, the number of days from the immediate study drug administration will be defined as 1 day.
- Complications of hepatobiliary disorders: Concurrent medical conditions summarized as hepatobiliary disorders by SOC.
- MAV: An abbreviation for markedly abnormal value.
- Overall hypoglycemia: Hypoglycemia reported as "Yes" for hypoglycemic symptoms and asymptomatic hypoglycemia.
- Asymptomatic hypoglycemia: Hypoglycemia with an evaluable self-monitoring blood glucose value (i.e., non-missing and determined to be eligible based on "Handling Rules for Analysis Data") and a measured concentration of ≤70 mg/dL but determined to be not accompanied by symptoms of hypoglycemia at the measurement of that blood glucose value. The presence or absence of asymptomatic hypoglycemia will be determined for each blood glucose value measured.

## HANDLING OF TIME WINDOW

For each test, observation, and evaluation items, evaluable data (i.e., non-missing data and data determined to be eligible based on "Handling Rules for Analysis Data") will be handled according to the following rules.

The evaluable data within the acceptable window will be used. If more than one evaluable datum lies within the same acceptable window, the data whose test/observation/evaluation date is closest to the scheduled date will be used and, if there are two data equidistant to the scheduled date, the data obtained earlier will be used for efficacy endpoints and the data obtained later will be used for safety endpoints.

HbA1c

| HOAIC | | _ | Acceptabl | e Window | |
|---|---|---|---|---|---|
| Visit | Scheduled Study Day | Study Day | Follow-up Day<br>for Treatment<br>Period I | Study Day for<br>Treatment<br>Period II | Follow-up Day<br>for SYR-472<br>25 mg Tablet |
| Week -6 | Study Day: -42 | -49 to -29 | | | |
| Week -2 | Study Day: -14 | -28 to -8 | | | |
| Week 0 | Study Day: 1 | -7 to 1 | | | |
| Week 2 | Study Day: 15 | 2 to 22 | ~ 20 | ~ 1 | |
| Week 4 | Study Day: 29 | 23 to 42 | ~ 20 | ~ 1 | |
| Week 8 | Study Day: 57 | 43 to 70 | ~ 20 | ~ 1 | |
| Week 12 | Study Day: 85 | 71 to 98 | ~ 20 | ~ 1 | |
| Week 16 | Study Day: 113 | 99 to 126 | | 2 ~ | ~ 20 |
| Week 20 | Study Day: 141 | 127 to 154 | | 2 ~ | ~ 20 |
| Week 24 | Study Day: 169 | 155 to 182 | | 2 ~ | ~ 20 |
| Week 28 | Study Day: 197 | 183 to 210 | | 2 ~ | ~ 20 |
| Week 32 | Study Day: 225 | 211 to 238 | | 2 ~ | ~ 20 |
| Week 36 | Study Day: 253 | 239 to 266 | | 2 ~ | ~ 20 |
| Week 40 | Study Day: 281 | 267 to 294 | | 2 ~ | ~ 20 |
| Week 44 | Study Day: 309 | 295 to 322 | | 2 ~ | ~ 20 |
| Week 48 | Study Day: 337 | 323 to 350 | | 2 ~ | ~ 20 |
| Week 52 | Study Day: 365 | 351 to 378 | | 2 ~ | ~ 20 |
| At the End of<br>Treatment Period I | Follow-up Day for<br>Treatment Period I: 7 | 2 ~ | ~ 20 | ~ 1 | |
| At the End of<br>Treatment Period II | Follow-up Day for SYR-472 25 mg Tablet: 7 | | | 2~* | ~ 20 |

<sup>\*:</sup> At the end of Treatment Period II, "Study Day for Treatment Period II" will be assumed to be "Study Day for SYR-472 25 mg tablet."

Fasting blood glucose

| rasting blood gi | | Acceptable Window | | | |
|---|---|---|---|---|---|
| Visit | Scheduled Study Day | Study Day | Follow-up Day<br>for Treatment<br>Period I | Study Day for<br>Treatment<br>Period II | Follow-up Day<br>for SYR-472<br>25 mg Tablet |
| Week -6 | Study Day: -42 | -49 to -22 | | | |
| Week 0 | Study Day: 1 | -21 to 1 | | | |
| Week 2 | Study Day: 15 | 2 to 22 | ~ 20 | ~ 1 | |
| Week 4 | Study Day: 29 | 23 to 42 | ~ 20 | ~ 1 | |

| | | Acceptable Window | | | |
|---|---|---|---|---|---|
| Visit | Scheduled Study Day | Study Day | Follow-up Day<br>for Treatment<br>Period I | Study Day for<br>Treatment<br>Period II | Follow-up Day<br>for SYR-472<br>25 mg Tablet |
| Week 8 | Study Day: 57 | 43 to 70 | ~ 20 | ~ 1 | |
| Week 12 | Study Day: 85 | 71 to 98 | ~ 20 | ~ 1 | |
| Week 16 | Study Day: 113 | 99 to 126 | | 2 ~ | ~ 20 |
| Week 20 | Study Day: 141 | 127 to 154 | | 2 ~ | ~ 20 |
| Week 24 | Study Day: 169 | 155 to 182 | | 2 ~ | ~ 20 |
| Week 28 | Study Day: 197 | 183 to 210 | | 2 ~ | ~ 20 |
| Week 32 | Study Day: 225 | 211 to 238 | | 2 ~ | ~ 20 |
| Week 36 | Study Day: 253 | 239 to 266 | | 2 ~ | ~ 20 |
| Week 40 | Study Day: 281 | 267 to 294 | | 2 ~ | ~ 20 |
| Week 44 | Study Day: 309 | 295 to 322 | | 2 ~ | ~ 20 |
| Week 48 | Study Day: 337 | 323 to 350 | | 2 ~ | ~ 20 |
| Week 52 | Study Day: 365 | 351 to 378 | | 2 ~ | ~ 20 |
| Week 54 | Follow-up Day for SYR-472 25 mg Tablet: 21 | | | | 21 to 28 |
| At the End of<br>Treatment Period I | Follow-up Day for<br>Treatment Period I: 7 | 2 ~ | ~ 20 | ~ 1 | |
| At the End of<br>Treatment Period II | Follow-up Day for SYR-472 25 mg Tablet: 7 | | | 2 ~ * | ~ 20 |

<sup>\*:</sup> At the end of Treatment Period II, "Study Day for Treatment Period II" will be assumed to be "Study Day for SYR-472 25 mg tablet."

Glycoalbumin

| | | Acceptable Window | | | |
|---|---|---|---|---|---|
| Visit | Scheduled Study Day | Study Day | Follow-up Day<br>for Treatment<br>Period I | Study Day for<br>Treatment<br>Period II | Follow-up Day<br>for SYR-472<br>25 mg Tablet |
| Week -6 | Study Day: -42 | -49 to -29 | | | |
| Week -2 | Study Day: -14 | -28 to -8 | | | |
| Week 0 | Study Day: 1 | -7 to 1 | | | |
| Week 2 | Study Day: 15 | 2 to 22 | ~ 20 | ~ 1 | |
| Week 4 | Study Day: 29 | 23 to 42 | ~ 20 | ~ 1 | |
| Week 8 | Study Day: 57 | 43 to 70 | ~ 20 | ~ 1 | |
| Week 12 | Study Day: 85 | 71 to 98 | ~ 20 | ~ 1 | |
| Week 16 | Study Day: 113 | 99 to 126 | | 2 ~ | ~ 20 |

| | | Acceptable Window | | | |
|---|---|---|---|---|---|
| Visit | Scheduled Study Day | Study Day | Follow-up Day<br>for Treatment<br>Period I | Study Day for<br>Treatment<br>Period II | Follow-up Day<br>for SYR-472<br>25 mg Tablet |
| Week 20 | Study Day: 141 | 127 to 154 | | 2 ~ | ~ 20 |
| Week 24 | Study Day: 169 | 155 to 182 | | 2 ~ | ~ 20 |
| Week 28 | Study Day: 197 | 183 to 210 | | 2 ~ | ~ 20 |
| Week 32 | Study Day: 225 | 211 to 238 | | 2 ~ | ~ 20 |
| Week 36 | Study Day: 253 | 239 to 266 | | 2 ~ | ~ 20 |
| Week 40 | Study Day: 281 | 267 to 294 | | 2 ~ | ~ 20 |
| Week 44 | Study Day: 309 | 295 to 322 | | 2 ~ | ~ 20 |
| Week 48 | Study Day: 337 | 323 to 350 | | 2 ~ | ~ 20 |
| Week 52 | Study Day: 365 | 351 to 378 | | 2 ~ | ~ 20 |
| Week 54 | Follow-up Day for<br>SYR-472 25 mg Tablet: 21 | | | | 21 to 28 |
| At the End of<br>Treatment Period I | Follow-up Day for<br>Treatment Period I: 7 | 2 ~ | ~ 20 | ~ 1 | |
| At the End of<br>Treatment Period II | Follow-up Day for SYR-472 25 mg Tablet: 7 | | | 2 ~ * | ~ 20 |

<sup>\*:</sup> At the end of Treatment Period II, "Study Day for Treatment Period II" will be assumed to be "Study Day for SYR-472 25 mg tablet."

Fasting C-peptide

| | | Acceptable Window | | | |
|---|---|---|---|---|---|
| Visit | Scheduled Study Day | Study Day | Follow-up Day<br>for Treatment<br>Period I | Study Day for<br>Treatment<br>Period II | Follow-up Day<br>for SYR-472<br>25 mg Tablet |
| Week -6 | Study Day: -42 | -49 to -29 | | | |
| Week -2 | Study Day: -14 | -28 to -8 | | | |
| Week 0 | Study Day: 1 | -7 to 1 | | | |
| Week 2 | Study Day: 15 | 2 to 22 | ~ 20 | ~ 1 | |
| Week 4 | Study Day: 29 | 23 to 42 | ~ 20 | ~ 1 | |
| Week 8 | Study Day: 57 | 43 to 70 | ~ 20 | ~ 1 | |
| Week 12 | Study Day: 85 | 71 to 98 | ~ 20 | ~ 1 | |
| Week 24 | Study Day: 169 | 99 to 210 | | 2 ~ | ~ 20 |
| Week 36 | Study Day: 253 | 211 to 308 | | 2 ~ | ~ 20 |
| Week 52 | Study Day: 365 | 309 to 378 | | 2 ~ | ~ 20 |
| Week 54 | Follow-up Day for SYR-472 25 mg Tablet: 21 | | | | 21 to 28 |

| | | Acceptable Window | | | |
|---|---|---|---|---|---|
| Visit | Scheduled Study Day | Study Day | Follow-up Day<br>for Treatment<br>Period I | Study Day for<br>Treatment<br>Period II | Follow-up Day<br>for SYR-472<br>25 mg Tablet |
| At the End of<br>Treatment Period I | Follow-up Day for<br>Treatment Period I: 7 | 2 ~ | ~ 20 | ~ 1 | |
| At the End of<br>Treatment Period II | Follow-up Day for SYR-472 25 mg Tablet: 7 | | | 2 ~ * | ~ 20 |

<sup>\*:</sup> At the end of Treatment Period II, "Study Day for Treatment Period II" will be assumed to be "Study Day for SYR-472 25 mg tablet."

Fasting glucagon, DPP-4 activity

| 1 asting gracagor | | Acceptable Window | | | |
|---|---|---|---|---|---|
| Visit | Scheduled Study Day | Study Day | Follow-up Day<br>for Treatment<br>Period I | Study Day for<br>Treatment<br>Period II | Follow-up Day<br>for SYR-472<br>25 mg Tablet |
| Week 0 | Study Day: 1 | -49 to 1 | | | |
| Week 2 | Study Day: 15 | 2 to 22 | ~ 20 | ~ 1 | |
| Week 4 | Study Day: 29 | 23 to 42 | ~ 20 | ~ 1 | |
| Week 8 | Study Day: 57 | 43 to 70 | ~ 20 | ~ 1 | |
| Week 12 | Study Day: 85 | 71 to 98 | ~ 20 | ~ 1 | |
| Week 24 | Study Day: 169 | 99 to 210 | | 2 ~ | ~ 20 |
| Week 36 | Study Day: 253 | 211 to 308 | | 2 ~ | ~ 20 |
| Week 52 | Study Day: 365 | 309 to 378 | | 2 ~ | ~ 20 |
| Week 54 | Follow-up Day for SYR-472 25 mg Tablet: 21 | | | | 21 to 28 |
| At the End of<br>Treatment Period I | Follow-up Day for<br>Treatment Period I: 7 | 2 ~ | ~ 20 | ~ 1 | |
| At the End of<br>Treatment Period II | Follow-up Day for SYR-472 25 mg Tablet: 7 | | | 2 ~ * | ~ 20 |

<sup>\*:</sup> At the end of Treatment Period II, "Study Day for Treatment Period II" will be assumed to be "Study Day for SYR-472 25 mg tablet."

Weight, BMI

| | | Acceptable Window | | | |
|---|---|---|---|---|---|
| Visit | Scheduled Study Day | Study Day | Follow-up Day<br>for Treatment<br>Period I | Study Day for<br>Treatment<br>Period II | Follow-up Day<br>for SYR-472<br>25 mg Tablet |
| Week -6 | Study Day: -42 | -49 to -29 | | | |
| Week -2 | Study Day: -14 | -28 to -8 | | | |
| Week 0 | Study Day: 1 | -7 to 1 | | | |
| Week 2 | Study Day: 15 | 2 to 22 | ~ 20 | ~ 1 | |

| | | Acceptable Window | | | |
|---|---|---|---|---|---|
| Visit | Scheduled Study Day | Study Day | Follow-up Day<br>for Treatment<br>Period I | Study Day for<br>Treatment<br>Period II | Follow-up Day<br>for SYR-472<br>25 mg Tablet |
| Week 4 | Study Day: 29 | 23 to 42 | ~ 20 | ~ 1 | |
| Week 8 | Study Day: 57 | 43 to 70 | ~ 20 | ~ 1 | |
| Week 12 | Study Day: 85 | 71 to 98 | ~ 20 | ~ 1 | |
| Week 16 | Study Day: 113 | 99 to 126 | | 2 ~ | ~ 20 |
| Week 20 | Study Day: 141 | 127 to 154 | | 2 ~ | ~ 20 |
| Week 24 | Study Day: 169 | 155 to 182 | | 2 ~ | ~ 20 |
| Week 28 | Study Day: 197 | 183 to 210 | | 2 ~ | ~ 20 |
| Week 32 | Study Day: 225 | 211 to 238 | | 2 ~ | ~ 20 |
| Week 36 | Study Day: 253 | 239 to 266 | | 2 ~ | ~ 20 |
| Week 40 | Study Day: 281 | 267 to 294 | | 2 ~ | ~ 20 |
| Week 44 | Study Day: 309 | 295 to 322 | | 2 ~ | ~ 20 |
| Week 48 | Study Day: 337 | 323 to 350 | | 2 ~ | ~ 20 |
| Week 52 | Study Day: 365 | 351 to 378 | | 2 ~ | ~ 20 |
| Week 54 | Follow-up Day for<br>SYR-472 25 mg Tablet: 21 | | | | 21 to 28 |
| At the End of<br>Treatment Period I | Follow-up Day for<br>Treatment Period I: 7 | 2 ~ | ~ 20 | ~ 1 | |
| At the End of<br>Treatment Period II | Follow-up Day for SYR-472 25 mg Tablet: 7 | | | 2 ~ * | ~ 20 |

<sup>\*:</sup> At the end of Treatment Period II, "Study Day for Treatment Period II" will be assumed to be "Study Day for SYR-472 25 mg tablet."

Vital signs, laboratory test, creatinine clearance, eGFR

| | | Acceptable Window | | | |
|---|---|---|---|---|---|
| Visit | Scheduled Study Day | Study Day | Follow-up Day<br>for Treatment<br>Period I | Study Day for<br>Treatment<br>Period II | Follow-up Day<br>for SYR-472<br>25 mg Tablet |
| Week -6 | Study Day: -42 | -49 to -29 | | | |
| Week -2 | Study Day: -14 | -28 to -8 | | | |
| Week 0 | Study Day: 1 | -7 to 1 | | | |
| Week 2 | Study Day: 15 | 2 to 22 | ~ 20 | ~ 1 | |
| Week 4 | Study Day: 29 | 23 to 42 | ~ 20 | ~ 1 | |
| Week 8 | Study Day: 57 | 43 to 70 | ~ 20 | ~ 1 | |
| Week 12 | Study Day: 85 | 71 to 98 | ~ 20 | ~ 1 | |

| | | | Acceptabl | Acceptable Window | |
|---|---|---|---|---|---|
| Visit | Scheduled Study Day | Study Day | Follow-up Day<br>for Treatment<br>Period I | Study Day for<br>Treatment<br>Period II | Follow-up Day<br>for SYR-472<br>25 mg Tablet |
| Week 16 | Study Day: 113 | 99 to 126 | | 2 ~ | ~ 20 |
| Week 20 | Study Day: 141 | 127 to 154 | | 2 ~ | ~ 20 |
| Week 24 | Study Day: 169 | 155 to 182 | | 2 ~ | ~ 20 |
| Week 28 | Study Day: 197 | 183 to 210 | | 2 ~ | ~ 20 |
| Week 32 | Study Day: 225 | 211 to 238 | | 2 ~ | ~ 20 |
| Week 36 | Study Day: 253 | 239 to 266 | | 2 ~ | ~ 20 |
| Week 40 | Study Day: 281 | 267 to 294 | | 2 ~ | ~ 20 |
| Week 44 | Study Day: 309 | 295 to 322 | | 2 ~ | ~ 20 |
| Week 48 | Study Day: 337 | 323 to 350 | | 2 ~ | ~ 20 |
| Week 52 | Study Day: 365 | 351 to 378 | | 2 ~ | ~ 20 |
| Week 54 | Follow-up Day for<br>SYR-472 25 mg Tablet: 21 | | | | 21 to 28 |

12-lead ECG

| | | Acceptable Window | | | |
|---|---|---|---|---|---|
| Visit | Scheduled Study Day | Study Day | Follow-up Day<br>for Treatment<br>Period I | Study Day for<br>Treatment<br>Period II | Follow-up Day<br>for SYR-472<br>25 mg Tablet |
| Week -6 | Study Day: -42 | -49 to -22 | | | |
| Week 0 | Study Day: 1 | -21 to 1 | | | |
| Week 4 | Study Day: 29 | 2 to 56 | ~ 20 | ~ 1 | |
| Week 12 | Study Day: 85 | 57 to 98 | ~ 20 | ~ 1 | |
| Week 24 | Study Day: 169 | 99 to 210 | | 2 ~ | ~ 20 |
| Week 36 | Study Day: 253 | 211 to 308 | | 2 ~ | ~ 20 |
| Week 52 | Study Day: 365 | 309 to 378 | | 2 ~ | ~ 20 |
| Week 54 | Follow-up Day for<br>SYR-472 25 mg Tablet: 21 | | | | 21 to 28 |

Plasma concentration of SYR-472Z

| | | Acceptable Window | | | |
|---|---|---|---|---|---|
| Visit | Scheduled Study Day | Study Day | Follow-up Day<br>for Treatment<br>Period I | Study Day for<br>Treatment<br>Period II | Follow-up Day<br>for SYR-472<br>25 mg Tablet |
| Week 4 | Study Day: 29 | 23 to 42 | ~ 20 | ~ 1 | |
| Week 12 | Study Day: 85 | 71 to 98 | ~ 20 | ~ 1 | |

#### OTHER HANDLING

• Creatinine clearance (mL/min): To be calculated using the following Cockcroft-Gault equation (rounded off to the nearest integer in both cases).

Male: ([140 – Age] × Weight [kg]) / (72 × Serum creatinine [mg/dL])

Female:  $0.85 \times ([140 - Age] \times Weight [kg]) / (72 \times Serum creatinine [mg/dL])$ 

Creatinine clearance will be calculated when the variables to be used for calculation are all evaluable and measured on the same day. The age will be calculated from the test dates of variables to be used for calculation and the date of birth.

• eGFR (mL/min/1.73 m<sup>2</sup>): To be calculated using the following equation (rounded off to the nearest integer in both cases).

Male:  $194 \times Serum$  creatinine  $(mg/dL)^{-1.094} \times Age^{-0.287}$ 

Female:  $194 \times \text{Serum creatinine (mg/dL)}^{-1.094} \times \text{Age}^{-0.287} \times 0.739$ 

The age will be calculated from the test dates of variables to be used for calculation and the date of birth.

- Duration of disease (months): Period from the onset time of type 2 diabetes until the time of informed consent.
- Duration of study drug exposure for Treatment Period I: Date of the last administration of the study drug for Treatment Period I – Date of the start of the study drug administration for Treatment Period I + 1
- Compliance with study drug for Treatment Period I: Number of study drug administrations for Treatment Period I / (Smallest integer of ≥ [(Date of the last administration of the study drug for Treatment Period I Date of the start of the study drug administration for Treatment Period I + 7) / 7]) × 100 (rounded off to the first decimal place)
- Duration of exposure to SYR-472 25 mg tablet: Date of the last administration of SYR-472
   25 mg tablet Date of the start of SYR-472 25 mg tablet + 1
- Compliance with SYR-472 25 mg tablet: Number of administrations of SYR-472 25 mg tablet / (Smallest integer of  $\geq$  [(Date of the last administration of SYR-472 25 mg tablet Date of the start of SYR-472 25 mg tablet + 7) / 7])  $\times$  100 (rounded off to the first decimal place)

#### 1 STUDY SUBJECTS, DEMOGRAPHICS, AND OTHER BASELINE CHARACTERISTICS

## 1.1 Disposition of Subjects

## 1.1.1 Study Information

Analysis set: All subjects who signed the informed consent form

Analysis variables: Date first subject signed the informed consent form

Date of last visit or contact, whichever comes later

MedDRA version
WHO Drug version

SAS version used for creating the datasets

Analysis methodology: The following analysis will be performed for the above analysis

variables.

(1) Display of the analysis variables

## 1.1.2 Disposition of All Subjects Who Were Not Randomized

Analysis set: All subjects who were not randomized

Analysis variables: Categories in brackets [ ] (hereinafter the same)

Age (years)  $[Min \le - < 65, 65 \le - \le Max]$ 

Sex [Male, Female]

Analysis methodology: The following analysis will be performed for the above analysis

variables.

(1) Frequency distributions for categorical variables and summary

statistics for continuous variables

## 1.1.3 Subject Eligibility

Analysis set: All subjects who signed the informed consent form

Analysis variables: Eligibility for randomization [Eligible, Not eligible]

Reason for not being randomized [Pretreatment event/Adverse

event, Significant protocol deviation, Lost to follow-up, Voluntary withdrawal, Study termination, Pregnancy, Did not meet inclusion criteria or did meet exclusion criteria,

Other]

Analysis methodology: The following analysis will be performed for the above analysis

variables.

When calculating percentages for the reasons for not being

randomized, the number of subjects who were not randomized will be used as the denominator.

(1) Frequency distribution

## 1.1.4 Number of Subjects Who Were Randomized by Site

Analysis set: All subjects who were randomized

Analysis variables: Eligibility for randomization [Eligible]

Stratum: Study site [Site numbers will be used as

categories]

Analysis methodology: The following analysis will be performed for the above analysis

variables for each stratum by each treatment group and in the

consolidated treatment groups.

(1) Frequency distribution

## 1.1.5 Disposition of Subjects

## 1.1.5.1 Disposition of Subjects in Treatment Period I

Analysis set: All subjects who were randomized

Analysis variables: Study drug administration status [Not treated]

Reason for not being treated [Pretreatment event/Adverse

event, Significant protocol deviation, Lost to follow-up, Voluntary withdrawal, Study termination, Pregnancy, Lack

of efficacy, Other]

Study drug administration status for [Treated, Not treated]

Treatment Period II

Reason for not being treated [Pretreatment event/Adverse

event, Significant protocol deviation, Lost to follow-up, Voluntary withdrawal, Study termination, Pregnancy, Lack

of efficacy, Other]

Analysis methodology: The following analysis will be performed for the above analysis

variables by each treatment group and in the consolidated treatment groups. When calculating percentages of the reasons for not being treated, the number of subjects who did not receive with the study

drug will be used as the denominator.

## (1) Frequency distribution

#### 1.1.5.2 Disposition of Subjects in the Entire Study

Analysis set: All subjects who were randomized

Analysis variables: Study drug administration status [Not treated]

Reason for not being treated [Pretreatment event/Adverse

event, Significant protocol deviation, Lost to follow-up, Voluntary withdrawal, Study termination, Pregnancy, Lack

of efficacy, Other]

Study drug completion status [Completed, Incompleted]

Reason for not being completed [Pretreatment event/Adverse

event, Significant protocol deviation, Lost to follow-up, Voluntary withdrawal, Study termination, Pregnancy, Lack

of efficacy, Other]

Completion status of the follow-up

period

[Completed, Incompleted]

Reason for not being completed [Pretreatment event/Adverse

event, Significant protocol deviation, Lost to follow-up, Voluntary withdrawal, Study termination, Pregnancy, Lack

of efficacy, Other]

Analysis methodology:

The following analysis will be performed for the above analysis variables by each treatment group and in the consolidated treatment groups. When calculating percentages of the reasons for not being treated, the number of subjects who did not receive the study drug will be used as the denominator. When calculating percentages of the reasons for not being completed, the number of subjects who did not complete the study drug/follow-up period will be used as the denominator.

(1) Frequency distribution

#### 1.1.6 Study Drug Completion Status

Analysis set: All subjects who were randomized

Analysis variables: Study drug completion status [Completed, Incompleted]

Reason for not being completed [Pretreatment event/Adverse

event, Significant protocol deviation, Lost to follow-up, Voluntary withdrawal, Study termination, Pregnancy, Lack

of efficacy, Other]

Categories: Number of study drug [0, 1-4, 5-8, 9-12, 13-24,

administrations 25-36, 37-48, 49-52,

53-Max]

Analysis methodology: The following analysis will be performed for the above analysis

variables by each treatment group and in the consolidated treatment

groups.

(1) Frequency distribution by number of study drug

administrations

#### 1.1.7 Protocol Deviations and Analysis Sets

### 1.1.7.1 Protocol Deviations

Analysis set: All subjects who were randomized

Analysis variables: Protocol deviations [Major GCP violations, Deviations of

protocol entry criteria, Deviations of discontinuation criteria, Deviations related to treatment procedure or dose, Deviations concerning excluded medication or therapy, Deviations to

avoid emergency risk, Other]

Analysis methodology: The following analysis will be performed for the above analysis

variables by each treatment group and in the consolidated treatment

groups.

Frequency distribution of subjects with protocol deviations will be provided for each deviation category above. A subject who has several deviations that can be classified into the same category will be counted once in each appropriate category (overlapped counting).

(1) Frequency distribution

#### 1.1.7.2 Analysis Sets

Analysis set: All subjects who were randomized

Analysis variables: Handling of subjects and subject [Categories are based on the

data in analysis sets specifications in "Handling

Rules for Analysis Data"]

Inclusion/Exclusion of analysis sets

Full analysis set [Included]
Per protocol set [Included]
Safety analysis set [Included]

Analysis methodology: The following analyses of (1) and (2) will be performed for the

above analysis variables by treatment group and the following

analysis of (3) will be performed by each treatment group and in the

consolidated treatment groups.

A subject who corresponds to several categories in (1) and (2) will be counted once in each appropriate category (overlapped counting).

(1) Frequency distributions concerning the handling of subjects in each analysis set

(2) Frequency distributions concerning the handling of subject data in each analysis set

(3) Frequency distributions concerning the number of subjects included in each analysis set

#### 1.2 Demographic and Other Baseline Characteristics

## 1.2.1 Distribution of Baseline Demographics

Analysis set: All subjects who were randomized

Analysis variables: Age (years)  $[Min \le - <65, 65 \le - \le Max]$ 

 $[Min \le - < 75, 75 \le - \le Max]$ 

Sex [Male, Female]

Height (cm)

Weight (kg) (Week 0)

BMI  $(kg/m^2)$  (Week 0) [Min  $\leq$  - <18.5, 18.5  $\leq$  - <25.0,

 $25.0 \le - < 30.0, 30.0 \le - \le Max$ 

Duration of disease (months)  $[Min \le - \le 24, 24 < - \le 60,$ 

 $60 < - \le 120, 120 < - \le Max$ 

Smoking status [Never smoked, Current

smoker, Ex-smoker]

Alcohol use [Yes, No]

Exercise therapy [Yes, No]

Hemodialysis [Yes (end-stage renal

failure), No (severe renal

impairment)]

[Yes, No]

Use of antidiabetic drugs (Week -6)

Rapid-acting insulin [Yes, No]

secretagogues

Details of rapid-acting insulin

secretagogues

Mitiglinide calcium hydrate [Yes]Repaglinide [Yes] $\alpha$ -glucosidase inhibitors [Yes, No]

Details of α-glucosidase inhibitors

Acarbose [Yes]
Miglitol [Yes]
Voglibose [Yes]

Insulin preparations [Yes, No]

Types of insulin preparations [Mixed, intermediate-acting,

Long-acting soluble]

Reason for concomitant use of

antidiabetic drugs being judged to

be appropriate

[Combination therapy is

expected to be more

effective, Development of

AEs due to dose increase is concerned, Maximum dose

has already been

administered, Other]

Creatinine (mg/dL) (Week 0) Male

Male  $[Min \le - \le 2.4, 2.4 < - \le Max]$ 

Female Female

 $[Min \le - \le 2.0, 2.0 \le - \le Max]$ 

Creatinine clearance (mL/min)

(Week 0)

eGFR (mL/min/1.73 m<sup>2</sup>) (Week 0)  $[Min \le -<15, 15 \le -<30,$ 

 $30 \le - \le Max$ 

HbA1c (%) (Week 0)  $[Min \le - <7.0, 7.0 \le - \le Max]$ 

[Min $\leq$  -  $\leq$ 8.0, 8.0 $\leq$  -  $\leq$ Max]

Fasting blood glucose (mg/dL)  $[Min \le -<130, 130 \le -<160,$ 

(Week 0)  $160 \le - \le Max$ 

Glycoalbumin (%) (Week 0)  $[Min \le - <24, 24 \le - \le Max]$ Fasting C-peptide (ng/mL) (Week 0)  $[Min \le - <1.0, 1.0 \le - <2.0,$ 

 $2.0 \le - \le Max$ 

Fasting glucagon (pg/mL) (Week 0) DPP-4 activity (nmol/min/mL)

(Week 0)

Analysis methodology: The following analysis will be performed for the above analysis

variables by each treatment group and in the consolidated treatment

groups. (1) Frequency distributions for categorical variables and

summary statistics for continuous variables

## 1.2.2 Medical History and Concurrent Medical Conditions

Analysis set: Safety analysis set

Analysis variables: Medical history

Concurrent medical conditions

Analysis methodology: The following analysis will be performed for the above analysis

variables by each treatment group and in the consolidated treatment

groups.

The analysis variables will be coded using MedDRA dictionary and will be summarized based on the SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

- (1) Frequency distributions for medical history (by SOC and PT)
- (2) Frequency distributions for concurrent medical conditions (by SOC and PT)

The frequency distributions will be provided according to the rules below:

[Number of subjects]

A subject with multiple occurrences of medical history or concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of medical history or concurrent medical condition within a PT will be counted only once in that PT.

## 1.2.3 Medication History and Concomitant Medications

Analysis set: Safety analysis set

Analysis variables: Medication history

Concomitant medications

Analysis methodology: The following analysis will be performed for the above analysis

variables by each treatment group and in the consolidated treatment

groups.

The analysis variables will be coded by use of WHO Drug and summarized based on Preferred Name, which will be sorted in decreasing frequency.

A subject who has been administered several medications with the same Preferred Name will be counted only once for that Preferred Name.

- (1) Frequency distributions for medication history
- (2) Frequency distributions for concomitant medications that were discontinued prior to the first dose of the study drug
- (3) Frequency distributions for concomitant medications that were ongoing at the first dose of the study drug and continued in the treatment period
- (4) Frequency distributions for concomitant medications that started after the first dose of the study drug
- (5) Frequency distributions for concomitant medications that were ongoing at the first dose of the study drug and continued in the treatment period, and concomitant medications that started after the first dose of the study drug

#### 1.2.4 Concomitant Antidiabetic Drugs Permitted in the Study

Analysis set: Full analysis set

Analysis variables: Newly added oral hypoglycemic drug [Yes, No]

in Treatment Period II (at Week 16

and thereafter)

Any change in antidiabetic drugs that [Yes, No]

are being used at Week -6 and will be concomitantly used during the study

period in Treatment Period II

Stratum: Types of antidiabetic drugs [Rapid-acting insulin

secretagogues,

α-glucosidase inhibitors,
Insulin preparations]

Analysis methodology:

The following analysis will be performed for the newly added oral hypoglycemic drug in Treatment Period II (at Week 16 and thereafter) in subjects who are not using any antidiabetic drug at Week -16 among the full analysis set by treatment group.

Also, the following analysis will be performed for any change in antidiabetic drugs that are being used at Week -6 and will be concomitantly used during the study period in Treatment Period II in subjects who are using antidiabetic drugs at Week -16 among the

Treatment Period II is the period from the start of the study drug administration for Treatment Period II until 20 days after the last administration of the study drug for Treatment Period II.

(1) Frequency distribution

full analysis set by treatment group.

#### 1.3 Measurement of Compliance Status for Treatment

#### 1.3.1 Study Drug Exposure and Compliance in the Treatment Period

| Analysis set: | Safety analysis set |
|---------------|---------------------|

Analysis variables: Number of study drug [1-12, 13-24, 25-36, 37-48,

administrations 49-52, 53-Max]

Number of study drug [1-4, 5-8, 9-12, 13-Max]

administrations in Treatment Period

I

Duration of study drug exposure in [1-28, 29-56, 57-84, 85-Max]

Treatment Period I (days)

Compliance with study drug for  $[Min \le - \le 50.0, 50.0 < - \le 70.0,$ 

Treatment Period I (%) 70.0< - \(\leq 90.0\), 90.0< - \(\leq \text{Max}\)

Number of administrations of [1-12, 13-24, 25-36, 37-48,

SYR-472 25 mg tablet 49-52, 53-Max]

Duration of exposure to SYR-472 [1-84, 85-168, 169-252,

25 mg tablet (days) 253-336, 337-364, 365-Max] Compliance with SYR-472 25 mg  $[Min \le - \le 50.0, 50.0 < - \le 70.0,$ 

tablet (%)  $70.0 < - \le 90.0, 90.0 < - \le \text{Max}$ 

Analysis methodology:

The following analysis will be performed for the above analysis variables by each treatment group and in the consolidated treatment groups.

(1) Frequency distributions for categorical variables and summary statistics for continuous variables

## 1.3.2 Compliance of Antidiabetic Drugs

Analysis set: Full analysis set

Analysis variables: Compliance with antidiabetic drugs [Fully complied (90% or

more), Almost complied (70% or more), Occasionally complied (50% or more), Rarely complied (less than

50%)]

Visits: Weeks -2, 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 or at

discontinuation, and 54

Analysis methodology: The following analysis will be performed for the above analysis

variables in subjects who are using antidiabetic drugs at Week -16 among the full analysis set by each treatment group and in the

consolidated treatment groups.

(1) Frequency distributions at each visit

#### 1.3.3 Compliance of Diet and/or Exercise Therapy

Analysis set: Full analysis set

Analysis variables: Compliance with diet [Fully complied (90% or

more), Almost complied

(70% or more), Occasionally complied (50% or more), Rarely complied (less than

50%)]

Compliance with exercise therapy [Fully complied (90% or

more), Almost complied

(70% or more), Occasionally complied (50% or more), Rarely complied (less than

50%)]

Visits: Weeks -2, 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 or at

discontinuation, and 54

Analysis methodology: The following analysis will be performed for the above analysis

variables by each treatment group and in the consolidated treatment

groups.

(1) Frequency distributions at each visit

#### 2 EFFICACY ANALYSIS

The "full analysis set" based on the specifications in the protocol and the "Handling Rules for Analysis Data" will be the main analysis set. For the sensitivity point of view, the "per protocol set" will be used for an analysis performed secondarily on the primary endpoint in order to examine the robustness of the results.

#### 2.1 Primary Endpoints and Analysis Methodology

## 2.1.1 Primary Analysis

Analysis set: Full analysis set

Analysis variables: Change in HbA1c at the end of Treatment Period I from Week 0 Analysis methodology: The population mean change in HbA1c at the end of Treatment

Period I from Week 0 will be compared between the SYR-472 25 mg/SYR-472 25 mg group and placebo/SYR-472 25 mg group based on an analysis of covariance (ANCOVA) model for the

change in HbA1c at the end of Treatment Period I from Week 0 with

factors of treatment group and HbA1c at Week 0.

The same ANCOVA model will be used to calculate the least square (LS) mean and the two-sided 95% confidence interval (CI) for each treatment group, as well as the intergroup difference in the LS mean between the treatment groups (SYR-472 25 mg/SYR-472 25 mg group – placebo/SYR-472 25 mg group) and the two-sided 95% CI.

#### 2.1.2 Secondary Analysis

Analysis set: Full analysis set

Per protocol set

Analysis variables: Change in HbA1c at the end of Treatment Period I from Week 0

Analysis methodology: The analysis (1) will be performed in the "full analysis set" and (2)

in the "per protocol set" for the above analysis variables.

(1) Summary statistics and the two-sided 95% CI for the mean will be calculated for each treatment group, as well as the intergroup difference in the mean between treatment groups (SYR-472 25 mg/SYR-472 25 mg group – placebo/SYR-472 25 mg group) and the two-sided 95% CI.

(2) In addition, the same analyses as 2.1.1 Primary Analysis and 2.1.2 Secondary Analysis (1) will be performed to evaluate the robustness of the results in terms of a sensitivity analysis.

#### 2.2 Secondary Endpoints and Analysis Methodology

## 2.2.1 HbA1c, Fasting Blood Glucose, Glycoalbumin

Analysis set: Full analysis set

Analysis variables: HbA1c

Fasting blood glucose

Glycoalbumin

Visits: HbA1c

Weeks -6, -2, 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, at the end of Treatment Period I, and at the end of Treatment Period II

Fasting blood glucose

Weeks -6, 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 54, at the end of Treatment Period I, and at the end of Treatment Period II

Glycoalbumin

Weeks -6, -2, 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 54, at the end of Treatment Period I, and at the end of Treatment Period II

Analysis methodology:

The following analyses (1) and (2) will be performed for the above analysis variables. Also, the following analysis (3) will be performed for HbA1c.

For the mean and standard deviation plot, a plot until Treatment Period I and a plot for the entire study will be created, respectively, but the plot for the entire period will not be output at Week 54 or at the end of Treatment Period I.

- (1) Summary statistics and the two-sided 95% CI for the mean will be calculated for each visit and the mean and standard deviation plot by treatment group will be prepared. Also, the intergroup difference in the mean between treatment groups (SYR-472 25 mg/SYR-472 25 mg group placebo/SYR-472 25 mg group) and the two-sided 95% CI will be calculated for each visit during the Screening and Treatment Period I.
- (2) The same analysis as the above (1) will be performed for changes from Week 0 at each visit after Treatment Period I.
- (3) For the proportions of subjects who achieved an HbA1c less than 6.0%, 7.0%, or 8.0% at the end of Treatment Period I and Treatment Period II, the proportions and the two-sided 95%

CIs will be calculated for each treatment group, and the intergroup difference in the proportions between treatment groups (SYR-472 25 mg/SYR-472 25 mg group – placebo/SYR-472 25 mg group) and the two-sided 95% CIs will be calculated at the end of Treatment Period I. In the analysis of each proportion, subjects who did not achieve the relevant target HbA1c at Week 0 will be included in the analysis.

#### 2.3 Other Endpoints and Analysis Methodology

#### 2.3.1 Fasting C-peptide, Fasting Glucagon, DPP-4 Activity, Weight

Analysis set: Full analysis set

Analysis variables: Fasting C-peptide

Fasting glucagon
DPP-4 activity

Weight

Visits: Fasting C-peptide

Weeks -6, -2, 0, 2, 4, 8, 12, 24, 36, 52, 54, at the end of Treatment

Period I, and at the end of Treatment Period II

Fasting glucagon, DPP-4 activity

Weeks 0, 2, 4, 8, 12, 24, 36, 52, 54, at the end of Treatment

Period I, and at the end of Treatment Period II

Weight

Weeks -6, -2, 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 54, at the end of Treatment Period I, and at the end of Treatment

Period II

Analysis methodology: The following analyses (1) and (2) will be performed for the above analysis variables.

For the mean and standard deviation plot, a plot until Treatment Period I and a plot for the entire study will be created respectively and the plot for the entire period will not be output at Week 54 and

at the end of Treatment Period I.

(1) Summary statistics and the two-sided 95% CI for the mean will be calculated for each visit and the mean and standard deviation plot by treatment group will be prepared. Also, the intergroup difference in the mean between treatment groups (SYR-472 25 mg/SYR-472 25 mg group – placebo/SYR-472

- 25 mg group) and the two-sided 95% CI will be calculated for each visit during the Screening and Treatment Period I.
- (2) The same analysis as the above (1) will be performed for changes from Week 0 at each visit after Treatment Period I (for DPP-4 activity, inhibition rate [100 × (Week 0 each visit after Treatment Period I) / Week 0, rounded off to the first decimal place]).

#### 2.4 Statistical and Analytical Issues

## 2.4.1 Adjustments for Covariates

See 2.1.1 Primary Analysis.

#### 2.4.2 Handling of Dropouts or Missing Data

Missing test results and ineligible data according to the "Handling Rules for Analysis Data" or the SAP will be excluded from statistical analyses and estimations.

#### 2.4.3 Interim Analysis and Data Monitoring

No interim analysis is planned.

#### 2.4.4 Multicenter Studies

Although this is a multicenter study, interactions between treatment and the study site will not be investigated since the target number of subjects per study site is not sufficiently large for meaningful analyses of the interactions.

#### 2.4.5 Multiple Comparisons/Multiplicity

The main focuses will be placed on the results of the primary analysis performed for the primary endpoint defined as "change in HbA1c at the end of Treatment Period I from Week 0" in the "full analysis set." Other analytical results will be interpreted to support the results of the primary endpoint or to explore the characteristics of efficacy of the study drug. These results will be considered one measure suggesting the trends or characteristics of efficacy. Thus, no adjustment for multiplicity will be performed.

## 2.4.6 Use of an "Efficacy Subset of Subjects"

To confirm the robustness of the primary analysis results for the primary endpoint for the sensitivity point of view, the same analysis as for the "full analysis set" will be performed secondarily in the "per protocol set."

#### 2.4.7 Active-Control Studies Intended to Show Equivalence or Non-inferiority

Not applicable.

#### 2.4.8 Examination of Subgroups

Analysis set: Full analysis set

Analysis variables: Change in HbA1c at the end of Treatment Period I from Week 0

Stratum: Age (years)  $[Min \le - <65, 65 \le - \le Max]$ 

Sex [Male, Female]

BMI  $(kg/m^2)$  (Week 0) [Min  $\leq$  -  $\leq$  25.0, 25.0  $\leq$  -

 $<30.0, 30.0 \le - \le Max$ 

Duration of disease (months)  $[Min \le - \le 120, 120 \le - \le Max]$ 

Medication history [Yes, No]

Hemodialysis [Yes (end-stage renal

failure), No (severe renal

impairment)]

Use of antidiabetic drugs (Week -6) [Yes, No]

Rapid-acting insulin secretagogues [Yes, No]

α-glucosidase inhibitors [Yes, No]

Insulin preparations [Yes, No]

eGFR (mL/min/1.73 m<sup>2</sup>) (Week 0)  $[Min \le -<15, 15 \le -\le Max]$ 

HbA1c (%) (Week 0)  $[Min \le - <7.0, 7.0 \le - \le Max]$ 

 $[Min \le - < 8.0, 8.0 \le - \le Max]$ 

Fasting blood glucose (mg/dL)  $[Min \le -<160, 160 \le -=Max]$ 

(Week 0)

Glycoalbumin (%) (Week 0)  $[Min \le - <24, 24 \le - \le Max]$ 

Fasting C-peptide (ng/mL)  $[Min \le - <2.0, 2.0 \le - \le Max]$ 

(Week 0)

Analysis methodology: The following analyses will be performed for the above analysis

variables.

(1) Summary statistics and the two-sided 95% CI for the mean will be calculated for each stratum by treatment group, as well as the intergroup difference in the mean between treatment groups (SYR-472 25 mg/SYR-472 25 mg group –

1 1 /OVD 470 05

placebo/SYR-472 25 mg group) and the two-sided 95% CI.

(2) The ANCOVA will be performed for each stratum with the change in HbA1c at the end of Treatment Period I from Week 0 as the response and with treatment group, stratum, and

interactions of treatment group and stratum as factors. The stratum will be included in the ANCOVA model as category variables based on the above category and analyzed.

## 2.5 Plasma Concentration of SYR-472Z

Analysis set: Full analysis set

Analysis variables: Plasma concentration of SYR-472Z

Stratum: Hemodialysis [Yes (end-stage renal

failure), No (severe renal

impairment)]

Visits: Weeks 4 and 12

Analysis methodology: Summary statistics will be calculated for the above analysis

variables for each visit in the SYR-472 25 mg/SYR-472 25 mg

group among the full analysis set.

The same analysis as the above will be performed for each stratum.

#### **3 SAFETY ANALYSIS**

#### 3.1 Treatment-Emergent Adverse Event

## 3.1.1 Overview of Treatment-Emergent Adverse Events

Analysis set: Safety analysis set

Analysis variables: TEAEs that occur before the start of the study drug for Treatment

Period II

TEAEs that occur after the start of SYR-472 25 mg tablet

Categories: Causality [Related, Not related]

Intensity [Mild, Moderate, Severe]

Analysis methodology: The following summaries will be provided for the above analysis

variables by treatment group.

In the analysis of TEAEs occurring after the start of SYR-472 25 mg tablet, subjects who received SYR-472 25 mg tablet in the safety analysis set will be included in the analyses and the summaries in the consolidated treatment groups will be also provided.

- (1) Overview of TEAEs
  - All TEAEs (number of events, number and percentage of subjects)
  - 2) Causal relationship between all TEAEs and study drug (number of events, number and percentage of subjects)
  - 3) Intensity of all TEAEs (number of events, number and percentage of subjects)
  - 4) TEAEs leading to study drug discontinuation (number of events, number and percentage of subjects)
  - 5) Serious TEAEs (number of events, number and percentage of subjects)
  - Causal relationship between serious TEAEs and study drug (number of events, number and percentage of subjects)
  - 7) Serious TEAEs leading to study drug discontinuation (number of events, number and percentage of subjects)
  - 8) TEAEs leading to death (number of events, number and percentage of subjects)

TEAEs will be counted according to the rules below:

[Number of subjects]

In the case of "summaries by causality"
 A subject with occurrences of TEAE in both categories (i.e.,

"Related" and "Not related") will be counted once in the "Related" category.

- In the case of "summaries by intensity"
   A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.
- In the case of summaries other than the above
   A subject with multiple occurrences of TEAE will be counted only once.

[Number of events]

For each summary, the total number of events will be calculated.

## 3.1.2 Displays of Treatment-Emergent Adverse Events

Analysis set: Safety analysis set

Analysis variables: TEAEs that occur before the start of the study drug for Treatment

Period II

TEAEs that occur after the start of SYR-472 25 mg tablet

Categories: Intensity [Mild, Moderate, Severe]

Time of onset (day)

TEAEs that occur before the

start of the study drug for

Treatment Period II

[1-28, 29-56, 57-Max]

[1-14, 15-28, 29-Max]

TEAEs that occur after the

start of SYR-472 25 mg

tablet

[1-84, 85-168, 169-252,

253-336, 337-Max]

[1-14, 15-28, 29-Max]

Number of days from the immediate [1, 2, 3, 4, 5, 6, 7, 8-Max]

study drug administration (days)

Analysis methodology: The following summaries will be provided for the above analysis

variables using frequency distributions by treatment group.

In the analysis of TEAEs occurring after the start of SYR-472 25 mg

tablet, subjects who received SYR-472 25 mg tablet in the safety analysis set will be included in the analyses and the summaries in

the consolidated treatment groups will be also provided concerning

(1) and (4).

TEAEs will be coded using MedDRA dictionary and will be summarized based on SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by SOC only or PT only.

- (1) All TEAEs by SOC and PT
- (2) All TEAEs by SOC
- (3) All TEAEs by PT
- (4) Drug-related TEAEs by SOC and PT
- (5) Intensity of all TEAEs by SOC and PT
- (6) Intensity of drug-related TEAEs by SOC and PT
- (7) TEAEs leading to study drug discontinuation by SOC and PT
- (8) Serious TEAEs by SOC and PT
- (9) All TEAEs by SOC and PT over time
- (10) Number of days from the immediate study drug administration for all TEAEs by SOC and PT
- (11) TEAEs whose incidence summarized by PT is 2% or higher (rounded off to the first decimal place) in either treatment group by SOC and PT
- (12) Intestinal obstruction-related TEAEs by SOC and PT
- (13) Acute pancreatitis-related TEAEs by SOC and PT
- (14) QT/QTc interval prolongation-related TEAEs by SOC and PT
- (15) Hypersensitivity-related TEAEs by SOC and PT
- (16) Cardiovascular TEAEs by SOC and PT
- (17) Pemphigoid TEAEs by SOC and PT
- (18) Renal impairment TEAEs by SOC and PT
- (19) Hypoglycemia-related TEAEs by SOC and PT

The frequency distribution and incidence will be provided according to the rules below:

#### [Number of subjects]

- In the case of "summaries by SOC and PT, by SOC, and by PT"
   A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages of TEAEs will be based on the number of subjects in the analysis set.
- In the case of "summaries of intensity by SOC and PT"

A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity. Percentages of TEAEs will be based on the number of subjects in the analysis set.

- In the case of "summaries by SOC and PT over time"

  A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT.

  When calculating percentages of TEAEs for each time interval, the number of subjects at risk (i.e., "subjects who either have an exposure in the study or have an occurrence of TEAE, during or after the corresponding time interval") will be used as the denominator. The number of subjects whose "onset of any one of the TEAEs is within the time interval" will be used as the numerator.
- In the case of "summaries of number of days from the immediate study drug administration" by SOC and PT
   A subject with a TEAE that occurs in more than one category of number of days is counted in all the categories that the TEAE occurs. For each category of number of days, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT. Percentages of TEAEs will be based on the number of subjects in the analysis set.

## 3.1.3 Subgroup Analysis of Treatment-Emergent Adverse Events

Analysis set: Safety analysis set

Analysis variables: TEAEs that occur before the start of the study drug for Treatment

Period II

TEAEs that occur after the start of SYR-472 25 mg tablet

Stratum: Age (years)  $[Min \le - <65, 65 \le - \le Max]$ 

 $[Min \le - < 75, 75 \le - \le Max]$ 

Hemodialysis [Yes (end-stage renal

failure), No (severe renal

impairment)]

Complications of hepatobiliary [Yes, No]

disorders

Use of antidiabetic drugs (Week -6) [Yes, No]

Rapid-acting insulin [Yes, No]

secretagogues

α-glucosidase inhibitors [Yes, No]Insulin preparations [Yes, No]

eGFR (mL/min/1.73 m<sup>2</sup>) (Week 0)  $[Min \le - <15, 15 \le - \le Max]$ 

Analysis methodology:

The following summaries will be provided for the above analysis variables using frequency distributions for each stratum by treatment group for TEAEs occurring before the start of the study drug for Treatment Period II and in the consolidated treatment groups for TEAEs occurring after the start of SYR-472 25 mg tablet.

In the analysis of TEAEs occurring after the start of SYR-472 25 mg tablet, subjects who received SYR-472 25 mg tablet in the safety analysis set will be included in the analyses. TEAEs will be coded using MedDRA dictionary and will be summarized based on SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

- (1) All TEAEs by SOC and PT
- (2) Drug-related TEAEs by SOC and PT

The frequency distributions will be provided according to the rules below:

[Number of subjects]

A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT.

#### 3.2 Pretreatment Event

#### 3.2.1 Display of Pretreatment Events

Analysis set: All subjects who signed the informed consent form

Analysis variables: PTE

Analysis methodology: The following summaries will be provided for the above analysis

variables using frequency distributions.

PTEs will be coded using MedDRA dictionary and will be summarized based on SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

(1) All PTEs by SOC and PT

## (2) Serious PTEs by SOC and PT

The frequency distributions will be provided according to the rules below:

[Number of subjects]

A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in that PT.

## 3.3 Clinical Laboratory Evaluations and Other Safety Endpoints

#### 3.3.1 Clinical Laboratory Evaluations

## 3.3.1.1 Hematology and Serum Chemistry

Analysis set: Safety analysis set

Analysis variables: Hematology

Red blood cells Reticulocytes White blood cells

HemoglobinHematocritPlateletsNeutrophilsLymphocytesMonocytes

Eosinophils Basophils MCV

MCH MCHC

Serum chemistry

ALT AST  $\gamma$ -GTP ALP

Total bilirubin Total protein
Albumin Creatinine
Amylase Lipase
Blood urea nitrogen Uric acid
Creatine kinase LDH

Total cholesterol Triglyceride

LDL cholesterol HDL cholesterol

High-sensitivity CRP K
Na Ca
Cl P

Fe Creatinine clearance

Categories: Adjudication results based on the normal reference ranges

[Low, Normal, High]

Visits: Weeks -6, -2, 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and

54

Analysis methodology:

The following analysis will be performed for the above analysis variables except for high-sensitivity CRP and creatinine clearance by treatment group. The following analyses of (1) to (2) will be performed for high-sensitivity CRP and creatinine clearance by treatment group.

When the analysis of MAV is performed, if both "upper" and "lower" criteria in the MAV Criteria are applicable to the same test item, the analysis will be performed for each criterion separately. See Appendix 2 of this SAP for the definitions of test items subject to this analysis and the MAV Criteria.

- (1) Summary statistics for each visit and summary statistics for change from Week 0 at each visit after Treatment Period I
- (2) Case plots
- (3) Shift tables showing adjudication results based on normal reference range at Week 0 and each visit after Treatment Period I
- (4) Frequency distributions for MAV before the start of the study drug administration for Treatment Period II and after the start of SYR-472 25 mg tablet

# 3.3.2 Vital Signs, Physical Examination, and Other Observation Items Related to Safety

## 3.3.2.1 Vital Signs

Analysis set: Safety analysis set

Analysis variables: Systolic blood pressure

Diastolic blood pressure

Pulse

Visits: Weeks -6, -2, 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and

54

Analysis methodology: The following analysis will be provided for the above analysis

variables by treatment group.

(1) Summary statistics for each visit and summary statistics for change from Week 0 at each visit after Treatment Period I

(2) Case plots

#### 3.3.2.2 12-lead ECG

Analysis set: Safety analysis set

Analysis variables: Heart rate

RR interval PR interval QRS interval

QT interval

QTcF interval

Findings of 12-lead ECG [Within normal limits,

Abnormal but not clinically significant, Abnormal and clinically significant]

Visits: Weeks -6, 0, 4, 12, 24, 36, 52, and 54

Analysis methodology: The following analyses of (1) to (3) will be performed for the above

analysis variables except for findings of 12-lead ECG by treatment

group.

The following analyses of (4) will be performed for findings of

12-lead ECG by treatment group.

When the analysis of MAV is performed, if both "upper" and "lower" criteria in the MAV Criteria are applicable to the same test

item, the analysis will be performed for each criterion separately.

See Appendix 2 of this SAP for the definitions of test items subject to this analysis and the MAV Criteria.

(1) Summary statistics for each visit and summary statistics for change from Week 0 at each visit after Treatment Period I

(2) Case plots

(3) Frequency distributions for MAV before the start of the study drug administration for Treatment Period II and after the start of SYR-472 25 mg tablet

(4) Shift tables showing at Week 0 and each visit after Treatment Period I

#### 3.3.2.3 Hypoglycemia

Analysis set: Safety analysis set

Analysis variables: Hypoglycemia that occurs after the start of the study drug

administration and before the start of the study drug for Treatment

Period II

Hypoglycemia that occurs after the start of SYR-472 25 mg tablet

Analysis methodology: The following summaries will be provided for the above analysis

variables using frequency distributions in subjects who

concomitantly received insulin preparations among the safety analysis set by treatment group.

In the analysis of hypoglycemia occurring after the start of SYR-472 25 mg tablet, subjects who concomitantly received insulin preparation and SYR-472 25 mg tablet in the safety analysis set will be included in the analyses.

- (1) All hypoglycemia
- (2) Severe hypoglycemia
- (3) Symptomatic hypoglycemia
- (4) Asymptomatic hypoglycemia
- (5) Probable symptomatic hypoglycemia
- (6) Relative hypoglycemia

The frequency distributions will be provided according to the rules below:

[Number of subjects]

A subject with multiple occurrences of hypoglycemia within the same classification will be counted only once in that classification.

[Number of events]

For each summary, the total number of events will be calculated.

## 4 SIGNIFICANCE LEVEL AND CONFIDENCE COEFFICIENT

• Significance level: 5% (two-sided tests)

• Confidence coefficient: 95% (two-sided)

# **History of Revision (version management)**

| Version | Date | F | Prepared/modified by | / | Comments |
|---|---|---|---|---|---|
| First Version | 16 April 2018 | | PPD | | Preparation of first version |
| Second Version | 12 June 2018 | | | | Preparation of second version |

## [Appendix 1] SYR-472-3003 Comparison Table for Changes

| Page | Existing Text | Revised Text | Rationale for Changes |
|---|---|---|---|
| 18 | 1.2.1 Distribution of Baseline Demographics | 1.2.1 Distribution of Baseline Demographics | Adjustment of descriptions and changes in |
| | Rapid-acting insulin secretagogues [Yes] | Rapid-acting insulin secretagogues [Yes, No] | the contents of distributions as a result of |
| | | Details of rapid-acting insulin secretagogues | reexamination of contents of distributions |
| | $\alpha$ -glucosidase inhibitors [Yes] | | |
| | | $\alpha$ -glucosidase inhibitors [Yes, No] | |
| | Insulin preparations [Yes] | Details of α-glucosidase inhibitors | |
| | Mixed [Yes] | | |
| | Intermediate-acting [Yes] | Insulin preparations [Yes, No] | |
| | Long-acting soluble [Yes] | Types of insulin preparations [Mixed, | |
| | | intermediate-acting, Long-acting soluble] | |
| 19 | 1.2.1 Distribution of Baseline Demographics | 1.2.1 Distribution of Baseline Demographics | Addition of distributions as a result of |
| | HbA1c (%) (Week 0) | HbA1c (%) (Week 0) | reexamination of contents of distributions |
| | [ $Min \le - < 8.0, 8.0 \le - \le Max$ ] | $[Min \le - <7.0, 7.0 \le - \le Max]$ | |
| | | [Min $\leq$ - $\leq$ 8.0, 8.0 $\leq$ - $\leq$ Max] | |
| 20 | 1.2.4 Concomitant Antidiabetic Drugs | 1.2.4 Concomitant Antidiabetic Drugs | Adjustment of descriptions to clarify the |
| | Permitted in the Study | Permitted in the Study | contents of distribution |
| | Any change in doses of antidiabetic drugs that | Any change in antidiabetic drugs that are | |
| | are being used at Week -6 and will be | being used at Week -6 and will be | |
| | concomitantly used during the study period in | concomitantly used during the study period in | |
| | Treatment Period II | Treatment Period II | |

| Page | Existing Text | Revised Text | Rationale for Changes |
|---|---|---|---|
| | Also, regarding the presence or absence of | Also, regarding the presence or absence of | |
| | any change in doses of antidiabetic drugs that | any change in antidiabetic drugs that are | |
| | are being used at Week -6 and will be | being used at Week -6 and will be | |
| | concomitantly used during the study period in | concomitantly used during the study period in | |
| | Treatment Period II, | Treatment Period II, | |
| 27 | 2.4.8 Examination of Subgroups | 2.4.8 Examination of Subgroups | Changes in the contents of distributions as a |
| | Duration of disease (months) | Duration of disease (months) | result of reexamination of categories at the |
| | $[Min \le - \le \underline{6}0, \underline{6}0 < - = Max]$ | $[Min \le - \le 120, 120 < - = Max]$ | blinded review |
| | Fasting C-peptide (ng/mL) | Fasting C-peptide (ng/mL) | |
| | $[Min \le - \le 1.0, 1.0 \le - \le 2.0, 2.0 \le - \le Max]$ | $[Min \le - <2.0, 2.0 \le - \le Max]$ | |
| 29 | 3.1.2 3.1.2 Displays of Treatment-Emergent | 3.1.2 3.1.2 Displays of Treatment-Emergent | Addition of distributions as a result of |
| | Adverse Events | Adverse Events | reexamination of contents of distributions |
| | | (19) Hypoglycemia-related TEAEs by SOC | |
| | | and PT | |